CLINICAL TRIAL: NCT01618292
Title: Cohort Study of Bowel Function Following Robotic-assisted Laparoscopic Sacrocolpopexy
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Jennifer Pagnillo, Patrick Culligan, MD, Atlantic Health System
Other Study IDs: R11-08-011
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Pelvic Organ Prolapse; Constipation; Bowel Dysfunction; Irritable Bowel Syndrome
Keywords: pelvic organ prolapse; constipation; bowel dysfunction; irritable bowel syndrome (IBS); CRADI-8; CRAIQ-7; splinting with defecation; excessive straining; bowel movements; fecal incontinence; bowel symptoms
MeSH Terms: conditions — Pelvic Organ Prolapse; Constipation; Intestinal Diseases; Irritable Bowel Syndrome; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Robotic-assisted sacrocolpopexy patients: Patients who underwent robotic-assisted laparoscopic sacrocolpopexy between January 2007 and August 2011.
  Interventions: Procedure: Robotic sacral colpopexy

INTERVENTIONS:
Procedure: Robotic sacral colpopexy — Patients who underwent robotic assisted sacral colpopexy for the treatment of pelvic organ prolapse
  Other Names: robotic-assisted laparoscopic sacral colpopexy

SUMMARY:
Compare changes in bowel function before, 6 months and one year after Robotic-assisted laparoscopic sacral colpopexy. Compare objective anatomic outcomes before, 6 months and one year after Robotic-assisted laparoscopic sacral colpopexy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent robotic assisted laparoscopic sacral colpopexy

Exclusion Criteria:

* Any other procedure for the treatment of pelvic organ prolapse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women suffering from pelvic organ prolapse who underwent a robotic assisted laparoscopic sacral colpopexy between January 2007 and August 2011.
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in bowel function | preoperatively, 6 months, and one year post-surgery
  -Patients completed a validated colo-rectal-anal distress inventory (CARDI-8) at all 3 intervals. Specific complaints of splinting with defecation, excessive straining/pain with bowel movements, incomplete bowel emptying/obstructive symptoms and fecal incontinence were addressed. In addition, patients completed a validated colorectal-anal impact questionnaire (CRAIQ-7) at all 3 intervals. The CRAIQ-7 addresses bowel symptoms and the extend of quality of life impingement

SECONDARY OUTCOMES:
Objective anatomic outcomes | preoperatively, 6 months, and one year after surgery
  The pelvic organ prolapse quantification system (POP-Q)- an objective, validated, standardized method of quantifying the degree of pelvic organ prolapse present was used at all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States